CLINICAL TRIAL: NCT02186756
Title: Biofeedback in Patients With Fibromyalgia - a Randomized Controlled Trial
Brief Title: A Randomized Controlled Trial to Evaluate the Effectiveness of Electromyography (EMG)-Biofeedback in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, PD Dr. Martin Weigl, MPH, PD, MD, MPH (Harvard University), Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PM-FMBFBack
Record Dates: First submitted 2014-07-02; First posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Complementary Therapies; Biofeedback; Randomized controlled trial; Relaxation Therapy
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMG-Biofeedback and Usual Care (Experimental): Patients in the intervention group started EMG-biofeedback training within three days after inclusion. In total 14 sessions of EMG-biofeedback training were applied. They started with three sessions of therapy in week 1-3 and had one session per week in week 4-8.
  Patients were encouraged to do a home exercise program, in which they consciously relaxed the muscle analogously to the biofeedback session for about 15 minutes per day. Additionally, they should try to apply the techniques in stressful situations, for example appointments at the dentist's.
  Interventions: Other: EMG-Biofeedback and Usual care
- Usual care (No Intervention): The patients in the control group had only two encounters with the therapist in the eight week interval. At these encounters pain was assessed by a visual analogue scale and their trapezius muscle activity was measured during 5 minutes analogously to the intervention group. However, afterwards they did not continue with muscle straining and relaxation.

INTERVENTIONS:
Other: EMG-Biofeedback and Usual care — Please refer to arm description
  Other Names: Schuhfried Biofeedback apparatus
  Arms: EMG-Biofeedback and Usual Care

SUMMARY:
The purpose of this study is to determine whether EMG-Biofeedback is effective in the treatment of Fibromyalgia.

DETAILED DESCRIPTION:
The objective of this randomized controlled trial is to evaluate the effectiveness of EMG-biofeedback in patients with Fibromyalgia. The assessors are blinded to the group assignment. There are three time points of assessment: before intervention, at the end of treatment (T1) and 3-months follow-up (T2). Patients are recruited from the waiting list of the Fibromyalgia day hospital program at the University Hospital Munich fulfilling the inclusion criteria. The intervention group is treated with 14 sessions of EMG-biofeedback during eight weeks in addition to usual care. The control group receives usual care only. The main specific aim is to assess the change in fibromyalgia specific health status.

ELIGIBILITY:
Inclusion Criteria:

* fibromyalgia according to the American Congress of Rheumatology (ACR)-criteria and the criteria.
* female gender
* age between 18 and 65
* cognitive ability and sufficient German language skills to fill in health status questionnaires
* signed informed consent

Exclusion Criteria:

* major medical disorders, i.e. cancer, chronic heart failure New York Heart Association (NYHA) IV or asthma requiring cortisone medication
* suffering from psychosis or major affective disorders
* substance abuse
* co-medication with opiates or benzodiazepine
* transmeridian flight in the last weeks
* shift-work
* gravity

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-04; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | Change from baseline to 3 months
  The primary outcome measure was the Fibromyalgia Impact Questionnaire (FIQ). The FIQ is a disease specific multidimensional self-administered instrument that covers the dimensions physical functioning (11 items), well-being (1 item), work situation (2 items), pain (1 item), fatigue /sleep (2 items), stiffness (2 items) and psychological symptoms (2 items). Scoring ranges from 0 to 80 with the latter number being the worst case. The FIQ Total Score gives a summary of patients' impairment and is recommended as a highly sensitive measure of change in Fibromyalgia treatment programs and clinical studies. In this study the validated German version was used.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | Change from baseline to End of Treatment (8 weeks after baseline)
Short-Form 36 (SF-36) | Change from baseline to End of treatment (8 weeks after baseline)
  The SF-36 is a widely used measure of health-related quality of life with 36 items. It yields an eight-scale profile of scores which are Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health.
Short-Form 36 (SF-36) | Change from baseline to 3 months
self-rated Patients' Global Clinical Impression of Change Score | End of Treatment (8 weeks after baseline)
  Change of health was directly measured by the self-rated Patients' Global Clinical Impression of Change Score, which is a validated measure of overall change compared with study onset, including six possible scores from "very much worse" (score 1) to "very much better" (score 6).
self-rated Patients' Global Clinical Impression of Change Score | 3 months
Beck Depression Inventory (BDI) | Change from baseline to End of treatment (8 weeks after baseline)
  This questionnaire was developed and validated for patients with depression and has been applied in clinical trials of patients with Fibromyalgia as well. It contains 21 items that assess the cognitive, affective and neurovegetative factors associated with depression.
Beck Depression Inventory (BDI) | Change from baseline to 3 months
Symptom Checklist 90 Revised (SCL-90-R) | Change from baseline to 3 Months
  the Symptom Checklist 90 Revised (SCL-90-R) was used for measuring psychological distress. It generates 9 specific scales, one additional unspecific scale and three general scores. The 9 dimensions of the scale are as follows: SCL 1 = somatization; SCL 2 = obsessive-compulsive symptoms; SCL 3 = interpersonal sensitivity; SCL 4 = depression; SCL 5 = anxiety; SCL 6 = hostility; SCL 7 = phobic anxiety; SCL 8 = paranoid ideation; SCL 9 = psychoticism. The Global Severity Index serves as a measure of psychological distress.
Tender Point Score | Change from baseline to End of treatment (8 weeks after baseline)
  It consists of a body diagram, where patients can rate the pain intensity at 24 locations of the front and the back side of the body. It allows calculating a total score for the whole body, as well as specific local scores.
Tender Point Score | Change from baseline to 3 months
Tender Point Count | Change from baseline to End of treatment (8 weeks after baseline)
  According to the Tender point manual the examiner applied discrete pressure of 4 kg/cm² to each of the 18 Fibromyalgia typical Tender Points. When the patients expressed pain, the tender point was considered positive.
Pressure Pain Threshold | Change from baseline to End of Treatment (8 weeks after baseline)
  For measuring the Pressure Pain Threshold, the assessor first searched for an induration with pressure pain in the trapezius muscle pars descendens on each side of the muscle. The palpated part of the muscle was always located above or on a line between the acromioclavicular joint and the spinous process of vertebrae C 7. These two structures also served as coordinates to write down the exact place of the palpated taut band. Second, using a Fischer dolorimeter with a stamp of 1 cm², the examiner applied vertical pressure to the selected point and successively augmented the pressure until the patient signalled pain. In this way, the pressure pain threshold was measured in kg/cm².

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Weigl, MD, MPH, Principal Investigator — Department of Orthopedics, Physical Medicine and Rehabilitation, University Hospital Munich, Ludwig Maximilians University Munich; Andreas Winkelmann, MD, Principal Investigator — Department of Orthopedics, Physical Medicine and Rehabilitation, University Hospital Munich, Ludwig Maximilians University Munich